CLINICAL TRIAL: NCT03648502
Title: Validation of "Montreal Cognitive Assessment (MoCA) and Addenbrooke's Cognitive Examination III (ACE-III) "as a Cognitive Screening Tools for the Hearing Impaired
Brief Title: Validation of Cognitive Screenings for the Hearing Impaired
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The corona virus pandemic_UK national lockdown
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 18/0306
Record Dates: First submitted 2018-08-02; First posted 2018-08-27 (Actual); Last update posted 2020-11-09 (Actual); Status verified 2020-11

CONDITIONS: Dementia; Hearing Loss; Auditory Processing Disorder
Keywords: dementia; hearing loss; auditory process
MeSH Terms: conditions — Dementia; Hearing Loss; Auditory Perceptual Disorders | interventions — Hearing Tests

STUDY DESIGN:
Intervention Model Description: 3 participants arms Diagnostic tools validation
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- dementia (D-HI) (Experimental): hearing impaired dementia
  Interventions: Diagnostic Test: Cognitive tests and hearing tests
- Mild cognitive impairment (MCI-HI) (Other): MCI with hearing loss
  Interventions: Diagnostic Test: Cognitive tests and hearing tests
- normal (N-HI) (Active Comparator): normal cognition with hearing loss
  Interventions: Diagnostic Test: Cognitive tests and hearing tests

INTERVENTIONS:
Diagnostic Test: Cognitive tests and hearing tests — Several cognitive and hearing (peripheral and (central) auditory process) tests

SUMMARY:
There are currently no cognitive tests that have been validated as screening tools for people with dementia and comorbid hearing loss. This is particularly important given the high prevalence of hearing impairment in older adults presenting to memory services and the risk of misdiagnosis of dementia in this population as outlined above.

Cognitive tests validated in hearing impaired populations will also be important as outcome tools for interventional research aiming to find out if treating hearing loss may reduce dementia risk in the longer term.

DETAILED DESCRIPTION:
Hearing loss is very prevalent in older population. This leads to further problems such as communication problem, isolation from the community and depression. Moreover, hearing impairment may potentially affect the patients' cognitive function as demonstrated in the above mentioned published papers.

Communication problems that arise from a hearing loss alone can also interfere with administration of cognitive test battery, as a previous study showed that re-administered of MMSE test with assistive listening device can immediately improve the test score among elderly (1).

Therefore, special adaptation of the cognitive test battery to address the needs of hearing impaired older adult is necessary. This is to ensure that the test result reflects the exact cognitive state of the older adult with hearing impairment, not effected by hearing loss.

Moreover, appropriate cut-off point scores for hearing impaired population should be identified for these new cognitive screening tools. This is to ensure appropriate referral for further diagnosis and prompt management for cognitive impairment/dementia among older adults with hearing loss.

In addition, since hearing loss can potentially lead to deterioration in patients' cognitive function over time (2). Follow up assessments of cognitive function among older adults with hearing impairment can determine the rate of deterioration in retrospective trial(2). This prospective trial follow up of cognitive function among hearing loss participants may uncover additional risk factors associated with the deterioration. Better understanding of these risk factors can potentially lead to further intervention in order to delay decline in patients' cognitive function.

ELIGIBILITY:
Inclusion Criteria:

* Age over 65 years
* Documented Hearing loss (currently wearing hearing aids and/or hearing testing with a hearing average of >/= 30dB HL in D-HI,MCI-HI group)

Exclusion criteria

* Uncorrected visual impairment; cognitive and/or physical disability(s) which prevent the performance of the written/drawing elements of the tests, in the opinion of the researcher.
* Severe to profound hearing loss (PTA >70dBHL)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 78 (Actual)
Dates: Start 2018-11-09 (Actual); Primary Completion 2020-03-13 (Actual); Study Completion 2020-03-13 (Actual)

PRIMARY OUTCOMES:
The adapted version Montreal Cognitive Assessment (MoCA) questionnaire total score among dementia/mild cognitive impairment/normal cognition group of hearing impaired older adult. | approximately 1 years (expected to recruit 30 participants for each group)
  The score will be used to calculate the appropriate cut-point score for differentiating each group of hearing impaired older adults.(total score ranging from 0-30 points with higher score indicate better cognitive function)
The adapted version Addenbrooke's Cognitive Examination III (ACE-III) questionnaire total score among dementia/mild cognitive impairment/normal cognition group of hearing impaired older adult. | approximately 1 years (expected to recruit 30 participants for each group)
  The score will be used to calculate the appropriate cut-point score for differentiating each group of hearing impaired older adults (total score ranging from 0-100 points with higher score indicate better cognitive function)

SECONDARY OUTCOMES:
Hearing handicap score from the Modified Amsterdam Inventory for Auditory Disability and Handicap (mAIAD) (total score ranging from 0-84 with higher score indicate smaller perceived hearing difficulty) | approximately 1 years (expected to recruit 30 participants for each group)
  The score from mAIAD and the hearing threshold from audiogram (in dB HL) along with the MoCA and ACE-III test scores will be used to determine what best predicts hearing handicap in the cognitively impaired population.

OTHER OUTCOMES:
Final cognitive status diagnosis (base on ICD-10 coding system; dichotomous outcome; code F00-F03 (dementia) or code ICD F06.7 (Mild cognitive impairment)) provided by an NHS memory service doctors at routine clinical care follow up session at 1 year. | 1 year follow up from initial recruitment
  The final cognitive status diagnosis of the population will be compared with hearing and cognitive outcome measures at baseline ie. the hearing threshold from audiogram (in dB HL)) and MoCA and ACE-III tests score and mAIAD questionnaire scores to determine what parameters best predict cognitive change in diagnosis from the baseline assessments in hearing impaired/cognitive impaired population.

CONTACTS AND LOCATIONS:
Overall Officials: Nattawan Utoomprurkporn, MD,Msc, Principal Investigator — University College, London
Locations (2):
- United Kingdom (2):
  - Royal National Throat Nose Ear Hospital, London
  - Camden and Islington NHS memory service, London

IPD SHARING:
Plan to Share IPD: No
only share within researchers team

REFERENCES:
- [Result] MacDonald AA, Joyson A, Lee R, Seymour DG, Soiza RL. The effect of hearing augmentation on cognitive assessment scales at admission to hospital. Am J Geriatr Psychiatry. 2012 Apr;20(4):355-61. doi: 10.1097/JGP.0b013e3182107e88. PMID 22434018
- [Result] Lin FR, Yaffe K, Xia J, Xue QL, Harris TB, Purchase-Helzner E, Satterfield S, Ayonayon HN, Ferrucci L, Simonsick EM; Health ABC Study Group. Hearing loss and cognitive decline in older adults. JAMA Intern Med. 2013 Feb 25;173(4):293-9. doi: 10.1001/jamainternmed.2013.1868. PMID 23337978